CLINICAL TRIAL: NCT00707434
Title: Continuous Glucose Monitoring Device Compared With Point-of-Care Glucose Testing in the ICU
Brief Title: Continuous Glucose Monitoring in Critically Ill
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Research administration changes.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2007-0616; NCI-2011-01085 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Results first posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Diabetes
Keywords: Continuous Glucose Monitor; Medtronic Guardian; Guardian® blood-sugar monitoring device; Glucose Monitoring; Critically Ill; ICU; Intensive Care Unit; Glycemic Excursions; Glucose Control; Glucose Testing; Hyperglycemia; Hypoglycemia; Insulin Infusion
MeSH Terms: conditions — Diabetes Mellitus; Critical Illness; Hyperglycemia; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Glucose Monitoring Device (Experimental): Continuous glucose monitoring in critically ill patients.
  Interventions: Device: Guardian® blood-sugar monitoring device

INTERVENTIONS:
Device: Guardian® blood-sugar monitoring device — The device has a small catheter that will be inserted subcutaneous tissue of the subject's abdomen or thigh set to continuously monitor glucose throughout the ICU stay for up to 15 days.
  Other Names: Continuous Glucose Monitor; Medtronic Guardian

SUMMARY:
The goal of this clinical research study is to learn if The Guardian® blood-sugar monitoring device can be used reliably in patients with high blood sugar who are receiving care in the ICU. Researchers will compare blood-sugar measurements from the study device with blood-sugar measurements from the standard "fingerstick" method of blood-sugar testing. This is being done to see if the new device can accurately measure blood sugar.

DETAILED DESCRIPTION:
The Study Device:

The Guardian® blood-sugar monitoring device is designed to automatically record blood sugar levels many times per hour, without requiring multiple fingersticks. It uses a blood sugar "sensor" (an electronic measuring device) that is about the size of a beeper. The sensor is attached to a small catheter that has a small needle in it. Once the catheter is inserted in the skin, the needle is removed right away.

Use of Study Device:

If you agree to take part in this study, while you are in the ICU, the catheter and needle part of the study device will be inserted under the skin of your abdomen or thigh. The device will automatically measure your blood sugar every 10 seconds so the data can be reviewed by the research staff. The needle will be removed right away. The catheter must be changed every 3 days (+/- 3 days) by the research staff. You will have the study device in place for 15 days (or until you leave the ICU, whichever comes first).

Standard Monitoring of Blood Sugar Levels:

While you are on study, your blood sugar will also be monitored according to the standard of care. This will be in the form of having your blood sugar checked by using a small needle to prick the tip of your finger every hour or more, as necessary.

The blood sugar measurements from the study device will not be used in any way to affect any decisions about your blood sugar monitoring or care.

Length of Study Participation:

After the study device is removed from your body for the last time (after 15 days or when you leave the ICU), you will be considered off study. If intolerable side effects occur, or an infection occurs that seems to have been caused by the study device, you will be taken off study early.

This is an investigational study. The study device is commercially available and FDA approved for monitoring blood sugar levels for outpatient (outside of the hospital) use. Using the device in patients who are in the hospital is considered experimental. At this time, it is only being used in this way in research.

Up to 60 patients will take part in this multicenter study. Up to 25 will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients in any of our University of Texas collaborative intensive care units.
2. Critically ill patients on an insulin infusion protocol

Exclusion Criteria:

1. Patients or their legal representatives who do not consent
2. Patients with large areas of skin affected so as not to allow implantation of device.
3. Patients < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-06; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naifa L. Busaidy, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (6):
- United States (6):
  - The University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Texas Health Science Center at Tyler, Tyler, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: June 12, 2008 to May 19, 2011. All recruitment was done at The University of Texas (UT) and UT MD Anderson Cancer Center.
Groups:
- Continuous Glucose Monitoring Device in ICU: Continuous glucose monitoring in critically ill patients throughout an intensive care unit (ICU) stay up to 15 days.
Period: Overall Study
Arm/Group | Continuous Glucose Monitoring Device in ICU
Started | 6
Completed | 5
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Continuous Glucose Monitoring in ICU: Continuous glucose monitoring in critically ill patients throughout an intensive care unit (ICU) stay up to 15 days.
Arm/Group | Continuous Glucose Monitoring in ICU
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 54 [47 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Mean Relative Difference in Patient Glucose Monitoring: Continuous Glucose Monitoring (CGM) Device as Compared With Point of Care (POC) Glucose Testing
Description: Mean relative difference will be calculated on a patient level assuming that at least 6 paired measurements will be collected from each patient.
  Outcome represents reliability of CGM device as compared with POC glucose testing where glucose values measured by POC will only be compared with the values read by the continuous glucose monitor sensor at the corresponding time points. The primary outcome for each patient is the mean relative difference defined as average of relative difference at each time point, where relative difference at each time point is calculated by taking difference in glucose values between CGM and POC and then divided by POC glucose value.
Time Frame: Continuously monitor patient's glucose throughout their ICU stay for up to 15 days.
Population: Study was terminated due to insufficient funding and data were not collected.
Arm/Group | Continuous Glucose Monitoring in ICU
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Participants monitored for up to 15 days or until leaving the ICU, whichever came first.
Arm/Group | Continuous Glucose Monitoring in ICU
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous Glucose Monitoring in ICU (N=6)
Bleeding at device insertion site (Injury, poisoning and procedural complications) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination led to small numbers of subjects analyzable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes